CLINICAL TRIAL: NCT03095690
Title: Determinants of Volumetric Bone Mineral Density at the Tibia and Radius and it's Relationship With Osteoporotic Fractures in Idiopathic Parkinson's Disease
Brief Title: Volumetric Bone Mineral Density and it's Relationship With Osteoporotic Fractures in Parkinson's Disease
Acronym: DOPPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2015-05
Record Dates: First submitted 2017-02-08; First posted 2017-03-30 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Osteoporosis; Parkinson; HR-pQCT; bone microstructure; fracture risk
MeSH Terms: conditions — Parkinson Disease; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idiopathic Parkinson's Disease patients (Other): High resolution peripheral scanner (HRpQCT).
  Interventions: Other: High resolution peripheral scanner (HRpQCT).

INTERVENTIONS:
Other: High resolution peripheral scanner (HRpQCT). — radius and tibia osteodensitometry measurement

SUMMARY:
Idiopathic Parkinson's disease (IPD) is the second most frequent neurodegenerative disease. Its association with osteroporosis and fragility fracture is now clearly demonstrated, but the determinants of this osteoporosis are yet to be explained. Our aim was to study factors associated with volumetric bone mineral density (vBMD) and bone microstructure at the tibia and radius in IPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease according to the criteria of the UKPDBB.
* Parkinson's disease of moderate severity (Index HOEHN and Yahr <5)
* Patient can respond to questionnaires, with or without help

Exclusion Criteria:

* Patients with active psychiatric illness preventing the realization of examinations
* Severe Parkinson's disease (Index HOEHN and Yahr ≥5 )
* Heavy-morbidity including heart failure NYHA> 3 or chronic respiratory failure, terminal or severe renal impairment known dialyzed
* Pregnancy

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Measurement of volumetric bone mineral density at the tibia and radius | 0 hour
  Measurement performed by High Resolution peripheral Quantitative Computed Tomography (HRpQCT)

CONTACTS AND LOCATIONS:
Overall Officials: Eric LESPESSAILLES, Ph, Principal Investigator — CHR d'ORLEANS
Locations (1):
- CHR d'ORLEANS, Orléans, France

IPD SHARING:
Plan to Share IPD: No